CLINICAL TRIAL: NCT00757588
Title: A Multicenter, Randomized, Double-Blind, Phase 3 Trial to Evaluate the Efficacy and Safety of Saxagliptin Added to Insulin Monotherapy or to Insulin in Combination With Metformin in Subjects With Type 2 Diabetes Who Have Inadequate Glycemic Control on Insulin Alone or on Insulin in Combination With Metformin
Brief Title: Safety and Efficacy of Saxagliptin Plus Insulin With or Without Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CV181-057; Eudract-2008-001089-10
Record Dates: First submitted 2008-09-22; First posted 2008-09-23 (Estimated); Results first posted 2011-12-13 (Estimated); Last update posted 2015-06-01 (Estimated); Status verified 2015-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — saxagliptin; Insulin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Saxagliptin, 5 mg + insulin (Experimental): Saxagliptin, 5 mg, plus insulin, administered to participants with Type 2 diabetes inadequately controlled with insulin alone or with insulin plus metformin
  Interventions: Drug: Saxagliptin, 5 mg + insulin
- Placebo + insulin (Placebo Comparator): Placebo administered to participants with Type 2 diabetes inadequately controlled with insulin alone or with insulin plus metformin
  Interventions: Drug: Placebo + insulin

INTERVENTIONS:
Drug: Saxagliptin, 5 mg + insulin — Saxagliptin, 5-mg tablets (plus stable insulin dose), given orally once daily (24 weeks short-term, 28 weeks long-term); participants stratified by use of stable metformin dose; flexible insulin dose (as needed for rescue)
  Other Names: BMS-477118
  Arms: Saxagliptin, 5 mg + insulin
Drug: Placebo + insulin — Placebo tablets given orally once daily for 24 weeks (short-term period)+ insulin with metformin
  Arms: Placebo + insulin

SUMMARY:
The purpose of this study is to compare the effects of saxagliptin with those of placebo as add-on therapy to insulin and insulin with metformin in improving glycemic control at 24 and 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus
* Must have been taking a stable dose of basal or premixed insulin for 8 weeks or longer prior to screening
* If taking metformin, must have been taking the same daily dose for 8 weeks or longer prior to screening
* Insulin type should be intermediate- or long-acting (basal) or premixed (premixed formulation may include short- or rapid-acting insulin as 1 component).
* Inadequate glycemic control (A1C of 7.5% to 11.0%, inclusive)
* Body mass index of 45 kg/m² or lower
* Fasting C-peptide level of 0.8 ng/mL or higher

Exclusion Criteria:

* Symptoms of poorly controlled diabetes, including but not limited to marked polyuria and polydipsia with greater than 10% weight loss during the last 3 months prior to screening or other signs and symptoms
* History of diabetic ketoacidosis or hyperosmolar nonketotic coma
* Women of childbearing potential unable or unwilling to use acceptable birth control
* Women who are pregnant or breastfeeding
* Active liver disease
* Anemia
* Chronic or repeated intermittent corticosteroid treatment (participants receiving stable doses of replacement corticosteroid (except dexamethasone) therapy may be enrolled)
* Use of short- or rapid-acting insulin
* Significant cardiovascular history defined as: myocardial infarction, coronary angioplasty or bypass graft, valvular disease or repair, unstable angina pectoris, transient ischemic attack, or cerebrovascular accident
* Congestive heart failure
* Unstable or rapidly progressing renal disease
* History of alcohol or drug abuse within the previous year
* History of hemoglobinopathies
* Unstable major psychiatric disorders
* Immunocompromised status

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2008-11; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (68):
- United States (16):
  - Clinical Research Advantage, Inc, Tempe, Arizona
  - Valley Research, Fresno, California
  - Torrance-Lomita Medical Center, Lomita, California
  - Diabetes Medical Center Of California, Northridge, California
  - Ritchken & First M.D.'S, San Diego, California
  - Encompass Clinical Research, Spring Valley, California
  - Central Florida Clinical Trials, Inc., Altamonte Springs, Florida
  - Family Care Associates Of Nw Florida, Chipley, Florida
  - Panhandle Family Care Assoc. & Coastal Palms Res. Grp Inc., Marianna, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Danny W. Jackson P.A., Rolling Fork, Mississippi
  - Southgate Medical Group, West Seneca, New York
  - Southeastern Research Associates, Inc., Taylors, South Carolina
  - Texas Center For Drug Development, Houston, Texas
  - Dgd Research, Inc., San Antonio, Texas
  - Aurora Advanced Healthcare, Milwaukee, Wisconsin
- Canada (9):
  - Local Institution, Calgary, Alberta
  - Local Institution, Vancouver, British Columbia
  - Local Institution, Bathurst, New Brunswick
  - Local Institution, London, Ontario
  - Local Institution, Charlottetown, Prince Edward Island
  - Local Institution, Gatineau, Quebec
  - Local Institution, Laval, Quebec
  - Local Institution, Sherbrooke, Quebec
  - Local Institution, Regina, Saskatchewan
- France (4):
  - Local Institution, Besançon
  - Local Institution, Montpellier
  - Local Institution, Nantes
  - Local Institution, Valenciennes
- Hungary (4):
  - Local Institution, Balatonfüred
  - Local Institution, Budapest
  - Local Institution, Szentes
  - Local Institution, Zalaegerszeg-Pozva
- India (5):
  - Local Institution, Indore, Madhya Pradesh
  - Local Institution, Hariyāna
  - Local Institution, Mumbai
  - Local Institution, Pune
  - Local Institution, Vellore
- Mexico (6):
  - Local Institution, Aguascalientes, Aguascalientes
  - Local Institution, Zapopan, Jal., Jalisco
  - Local Institution, Mexico City, Mexico City
  - Local Institution, Monterrey, Nuevo León
  - Local Institution, Monterrrey, Nuevo León
  - Local Institution, Veracruz, Veracruz
- Poland (9):
  - Local Institution, Elblag
  - Local Institution, Gdansk
  - Local Institution, Krakow
  - Local Institution, Lodz
  - Local Institution, Lublin
  - Local Institution, Sopot
  - Local Institution, Szczecin
  - Local Institution, Wroclaw
  - Local Institution, Zabrze
- Russia (5):
  - Local Institution, Kursk
  - Local Institution, Saint Petersburg
  - Local Institution, Saratov
  - Local Institution, Smolensk
  - Local Institution, Yaroslaval
- South Africa (5):
  - Local Institution, Parktown, Gauteng
  - Local Institution, Durban, KwaZulu-Natal
  - Local Institution, Umhlanga, KwaZulu-Natal
  - Local Institution, Goodwood, Western Cape
  - Local Institution, Tygerberg, Western Cape
- United Kingdom (5):
  - Local Institution, Middlesbrough, Cleveland
  - Local Institution, Salford, Greater Manchester
  - Local Institution, Newcastle upon Tyne, Tyne and Wear
  - Local Institution, Birmingham, West Midlands
  - Local Institution, Sheffield, Yorkshire

REFERENCES:
- [Derived] Perl S, Cook W, Wei C, Iqbal N, Hirshberg B. Saxagliptin Efficacy and Safety in Patients With Type 2 Diabetes and Moderate Renal Impairment. Diabetes Ther. 2016 Sep;7(3):527-35. doi: 10.1007/s13300-016-0184-9. Epub 2016 Jul 11. PMID 27402391
- [Derived] Cook W, Minervini G, Bryzinski B, Hirshberg B. Saxagliptin efficacy and safety in patients with type 2 diabetes mellitus stratified by cardiovascular disease history and cardiovascular risk factors: analysis of 3 clinical trials. Postgrad Med. 2014 Oct;126(6):19-32. doi: 10.3810/pgm.2014.10.2818. PMID 25414932
- [Derived] Barnett AH, Charbonnel B, Li J, Donovan M, Fleming D, Iqbal N. Saxagliptin add-on therapy to insulin with or without metformin for type 2 diabetes mellitus: 52-week safety and efficacy. Clin Drug Investig. 2013 Oct;33(10):707-17. doi: 10.1007/s40261-013-0107-8. PMID 23949898
- [Derived] Barnett AH, Charbonnel B, Donovan M, Fleming D, Chen R. Effect of saxagliptin as add-on therapy in patients with poorly controlled type 2 diabetes on insulin alone or insulin combined with metformin. Curr Med Res Opin. 2012 Apr;28(4):513-23. doi: 10.1185/03007995.2012.665046. Epub 2012 Mar 1. PMID 22313154
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of 455 participants randomized, 402 received treatment and completed the 24-week phase. Two participants were mistakenly identified as not completing the short-term (ST) treatment period, although they did. The discrepancy was identified after the ST phase database lock. In reality, 404 completed the ST phase.
Groups:
- Saxagliptin, 5 mg + Insulin: Saxagliptin, 5 mg, added to ongoing insulin with or without metformin therapy for up to 24 weeks in patients with type 2 diabetes
- Placebo + Insulin: Placebo added to ongoing insulin with metformin therapy for up to 24 weeks in patients with type 2 diabetes
Period: Period 1: Short-term (24-week) Phase
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Started | 304 | 151
Completed | 268 (Does not include 2 who completed Period 1 but were erroneously reported in the CSR as noncompleters.) | 134
Not Completed | 36 | 17
Not completed — Lack of Efficacy | 3 | 2
Not completed — Adverse Event | 6 | 3
Not completed — Withdrawal by Subject | 13 | 5
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 3 | 5
Not completed — Poor compliance or noncompliance | 5 | 1
Not completed — No longer meets study criteria | 5 | 0
Not completed — Other | 0 | 1
Period: Period 2: Long-term (52-week) Phase
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Started | 268 (270 participants completed short-term phase; 2 of these did not enter long-term phase.) | 134
Completed | 246 | 125
Not Completed | 22 | 9
Not completed — Lack of Efficacy | 1 | 0
Not completed — Adverse Event | 4 | 0
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Poor or noncompliance | 5 | 2
Not completed — Pregnancy | 1 | 0
Not completed — No longer meets study criteria | 5 | 4
Not completed — Other | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin | Total
Number analyzed (Participants) | 304 | 151 | 455
Age, Customized [Median (Full Range); unit: years] | 58 (9.43) [18 to 77] | 58 (9.27) [30 to 77] | 58 (9.37) [18 to 77]
Age, Customized [Number; unit: participants]
  Younger than 65 years | 233 | 118 | 351
  65 years to younger than 75 years | 65 | 30 | 95
  75 years and older | 6 | 3 | 9
Age, Customized [Mean (Standard Deviation); unit: Years] | 57.2 (9.43) | 57.3 (9.27) | 57.2 (9.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 184 | 83 | 267
  Male | 120 | 68 | 188
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 40 | 19 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 9 | 22
  White | 237 | 118 | 355
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 14 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change From Baseline in A1C Levels (Last Observation Carried Forward [LOCF])
Description: Change from baseline: post-pre. Adjusted for baseline (value and metformin use). ANCOVA model: difference between week t and baseline values=baseline values + treatment + metformin use
Time Frame: Baseline to Week 24
Population: Randomized participants who received at least 1 dose of double-blind study medication. Participants must also have had both a baseline and at least 1 postrandomization measurement in the 24- and 52-week periods.
Measure: Mean (Standard Error); unit: Percentage of change
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 300 | 149
Percentage of change | -0.73 (0.054) | -0.32 (0.074)
Statistical Analysis 1: Comparison: Saxagliptin, 5 mg + Insulin; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-0.59 to -0.24], Standard Error of Mean 0.089 — ANCOVA model: difference between week t and baseline values = baseline values + treatment + metformin use

2. Secondary Outcome: Change From Baseline in Postprandial Glucose (PPG) Area Under the Curve (AUC) Response to an Meal Tolerance Test (MTT)
Description: An MTT is a 2-part test that measures glucose and insulin levels after an overnight fast and before ingesting a meal consisting of a nutritional drink and power bar and again at prespecified times (30, 60, 120, and 180 minutes) after the start of ingestion of the meal
Time Frame: Baseline to Week 24
Measure: Mean (Standard Error); unit: mg*min/dL
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 258 | 122
mg*min/dL | -4548.5 (687.65) | -718.8 (981.63)
Statistical Analysis 1: Comparison: Saxagliptin, 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p = 0.0011, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -3829.8, 95% CI 2-sided [-6122.4 to -1537.1], Standard Error of Mean 1165.99 — ANCOVA model: difference between week t and baseline values = baseline values + treatment + metformin use

3. Secondary Outcome: Change From Baseline in 120-minute PPG Values During an MTT
Description: as for outcome 2
Time Frame: Baseline to Week 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 262 | 129
mg/dL | -27.2 (4.35) | -4.2 (6.08)
Statistical Analysis 1: Comparison: Saxagliptin, 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p = 0.0016, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -23.0, 95% CI 2-sided [-37.2 to -8.7], Standard Error of Mean 7.24 — ANCOVA model: difference between week t and baseline values = baseline values + treatment + metformin use

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose Values
Time Frame: Baseline to Week 24
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 300 | 149
mg/dL | -10.1 (2.87) | -6.1 (3.98)
Statistical Analysis 1: Comparison: Saxagliptin, 5 mg + Insulin vs Placebo + Insulin; Test type: Superiority or Other; p = 0.3958, ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -4.02, 95% CI 2-sided [-13.32 to 5.28], Standard Error of Mean 4.732 — ANCOVA model: difference between week t and baseline values = baseline values + treatment + metformin use

5. Secondary Outcome: Percentage of Participants Achieving a Therapeutic Glycemic Response
Description: Therapeutic glycemic response is defined as an A1C<7%. Significance was not interpreted with a p value.
Time Frame: Baseline to Week 24
Population: Randomized participants who received at least 1 dose of double-blind study medication. Participants must also have had both a baseline and at least 1 postrandomization measurement in the 24-week period.
Measure: Number; unit: Percentage of participants
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 300 | 149
Percentage of participants | 17.3 | 6.7

6. Secondary Outcome: Change From Baseline in Mean Total Daily Dose of Insulin (MTDDI) (LOCF)
Description: Based on information recorded in the participant's daily diary. The MTDDI was calculated at every visit using the values patients recorded since the last regularly scheduled visit (minimum of 80% of days with a value). At every visit, the MTDDI was compared with the participant's baseline MTDDI (measured during a 4-week lead-in period) to identify any changes in insulin use at that visit compared with insulin use at baseline.
Time Frame: Baseline to Week 24
Population: as for outcome 5
Measure: Mean (Standard Error); unit: Units
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 299 | 151
Units | 1.71 (0.704) | 5.01 (0.970)
Statistical Analysis 1: Comparison: Saxagliptin, 5 mg + Insulin; Test type: Superiority or Other; ANCOVA — Significance testing based on hierarchical testing. Primary and secondary endpoints are presented in order of testing; Adjusted mean difference for saxagliptin groups vs placebo in Week 24 (LOCF). Adjusted for baseline; Mean Difference (Final Values) = -3.3, 95% CI 2-sided [-5.6 to -1.1], Standard Error of Mean 1.16 — ANCOVA model: difference between week t and baseline values = baseline values + treatment + metformin use

7. Other Pre Specified Outcome: Number of Participants With Abnormal Changes From Baseline in Electrocardiogram (ECG) Results
Description: ECG abnormalities included those in nonspecific "other" categories (Other nonspecific ST/T, Other intraventricular conduction defect, Other, and Other rhythm abnormalities)and nonspecific findings, such as sinus bradycardia, sinus arrythmia, sinus tachycardia, poor R-wave progression, and ventricular premature contractions.
Time Frame: Baseline to Week 52
Population: Participants who had normal ECG findings at baseline and who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 153 | 75
Participants | 15 | 11

8. Other Pre Specified Outcome: Shift in Absolute Lymphocyte Counts From Baseline to Selected Visits (LOCF)
Description: Absolute lymphocyte count=value*10^3 c/uL
Time Frame: Baseline and Weeks 24 and 52
Population: All participants who received at least 1 dose of double-blind study medication.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 304 | 151
Participants
  Baseline <= 0.75; Week 24 <= 0.75 | 0 | 0
  Baseline <= 0.75; Week 24 >0.75- <= 5.00 | 0 | 2
  Baseline <= 0.75; Week 24 >5.00 | 0 | 0
  Baseline >0.75- <= 5.00; Week 24 <= 0.75 | 1 | 0
  Baseline >0.75- <= 5.00; Week 24 >0.75- <= 5.00 | 293 | 148
  Baseline >0.75- <= 5.00; Week 24 >5.00 | 1 | 0
  Baseline >5.00; Week 24 <= 0.75 | 0 | 0
  Baseline >5.00; Week 24 >0.75- <= 5.00 | 0 | 0
  Baseline >5.00; Week 24 >5.00 | 1 | 0
  Baseline <= 0.75; Week 52 <= 0.75 | 0 | 0
  Baseline <= 0.75; Week 52 >0.75- <= 5.00 | 0 | 2
  Baseline <= 0.75; Week 52 >5.00 | 0 | 0
  Baseline >0.75- <= 5.00; Week 52 <= 0.75 | 0 | 0
  Baseline >0.75- <= 5.00; Week 52 >0.75- <= 5.00 | 295 | 147
  Baseline >0.75- <= 5.00; Week 52 >5.00 | 0 | 1
  Baseline >5.00; Week 52 <= 0.75 | 0 | 0
  Baseline >5.00; Week 52 >0.75- <= 5.00 | 0 | 0
  Baseline >5.00; Week 52 >5.00 | 1 | 0

9. Other Pre Specified Outcome: Number of Participants With at Least 1 Adverse Event (AE), at Least 1 Treatment-related AE, Death as Outcome, at Least 1 Serious Adverse Event (SAE), at Least 1 Treatment-related SAE, Discontinuations Due to SAEs, and Discontinuations Due to AEs
Description: An AE is any new untoward medical occurrence or worsening of a preexisting medical condition that does not necessarily have a causal relationship with this treatment. An SAE is any untoward medical event that at any dose: results in death, persistent or significant disability/incapacity, or drug dependency or abuse; is life-threatening, an important medical event, or a congenital anomaly/birth defect; requires inpatient hospitalization; or prolongs existing hospitalization. Treatment-related=possibly, probably, or certainly related to and of unknown relationship to study treatment.
Time Frame: Baseline to Week 52, continuously
Population: All participants who received at least 1 dose of double-blind study medication.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 304 | 151
Participants
  At least 1 AE | 202 | 108
  At least 1 treatment-related AE | 56 | 34
  Deaths | 2 | 0
  At least 1 SAE | 25 | 13
  At least 1 treatment-related SAE | 3 | 0
  Discontinuations due to SAEs | 4 | 0
  Discontinuations due to AEs | 9 | 3

10. Other Pre Specified Outcome: Mean Changes From Baseline in Systolic and Diastolic Blood Pressure Readings
Time Frame: Baseline to Weeks 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, 44, and 52
Population: All participants who received at least 1 dose of double-blind study medication.
Measure: Number (95% Confidence Interval); unit: mm Hg
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 304 | 151
mm Hg
  Systolic blood pressure (Week 2) (n=294, 147) | -1.0 [-2.3 to 0.4] | 2.3 [-0.0 to 4.6]
  Systolic blood pressure (Week 4) (n=293, 144) | -1.2 [-2.6 to 0.2] | 0.0 [-2.3 to 2.4]
  Systolic blood pressure (Week 6) (n=280, 141) | -0.8 [-2.4 to 0.7] | 1.0 [-1.2 to 3.2]
  Systolic blood pressure (Week 8) (n=290, 142) | -0.8 [-2.4 to 0.8] | 2.4 [-0.2 to 4.9]
  Systolic blood pressure (Week 12) (n=286, 144) | -1.7 [-3.2 to -0.2] | 2.2 [0.0 to 4.3]
  Systolic blood pressure (Week 16) (n=278, 139) | -1.2 [-2.9 to 0.5] | 1.1 [-1.1 to 3.3]
  Systolic blood pressure (Week 20) (n=276, 137) | -0.6 [-2.0 to 0.9] | 1.3 [-1.0 to 3.7]
  Systolic blood pressure (Week 24) (n=273, 134) | -1.5 [-3.2 to 0.1] | -0.1 [-2.2 to 2.0]
  Systolic blood pressure (Week 28) (n=264, 132) | -1.4 [-3.0 to 0.1] | 1.8 [-0.6 to 4.2]
  Systolic blood pressure (Week 36) (n=261, 129) | -0.7 [-2.4 to 1.1] | 3.6 [1.2 to 6.0]
  Systolic blood pressure (Week 44) (n=250, 125) | -0.6 [-2.2 to 1.0] | 2.6 [0.4 to 4.8]
  Systolic blood pressure (Week 52) (n=246, 125) | 0.0 [-1.7 to 1.7] | 1.0 [-1.3 to 3.3]
  Diastolic blood pressure (Week 2) (n=294, 147) | 0.1 [-0.9 to 1.0] | 1.4 [-0.0 to 2.8]
  Diastolic blood pressure (Week 4) (n=293, 144) | 0.0 [-1.0 to 1.1] | 1.8 [0.4 to 3.2]
  Diastolic blood pressure (Week 6) (n=280, 141) | 0.0 [-1.0 to 1.1] | 0.3 [-1.1 to 1.8]
  Diastolic blood pressure (Week 8) (n=290, 142) | -0.5 [-1.5 to 0.4] | 2.1 [0.6 to 3.6]
  Diastolic blood pressure (Week 12) (n=286, 144) | -0.8 [-1.8 to 0.2] | 1.0 [-0.3 to 2.4]
  Diastolic blood pressure (Week 16) (n=278, 139) | -1.1 [-2.1 to -0.1] | 1.3 [-0.0 to 2.6]
  Diastolic blood pressure (Week 20) (n=276, 137) | -0.7 [-1.8 to 0.4] | 1.1 [-0.3 to 2.5]
  Diastolic blood pressure (Week 24) (n=273, 134) | -1.7 [-2.8 to -0.6] | 0.5 [-0.9 to 1.9]
  Diastolic blood pressure (Week 28) (n=264, 132) | -1.6 [-2.7 to -0.5] | 0.2 [-1.3 to 1.7]
  Diastolic blood pressure (Week 36) (n=261, 129) | -1.2 [-2.4 to 0.1] | 0.2 [-1.1 to 1.6]
  Diastolic blood pressure (Week 44) (n=250, 125) | -0.3 [-1.5 to 1.0] | 0.4 [-1.0 to 1.8]
  Diastolic blood pressure (Week 52) (n=246, 125) | -0.5 [-1.7 to 0.7] | 0.1 [-1.4 to 1.6]

11. Other Pre Specified Outcome: Mean Changes From Baseline in Heart Rate
Time Frame: Baseline to Weeks 2, 4, 6, 8, 12, 16, 20, 24, 28, 36, 44, and 52
Population: All participants who received at least 1 dose of double-blind study medication.
Measure: Number (95% Confidence Interval); unit: Beats per minute
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 304 | 151
Beats per minute
  Week 2 (n=294, 147) | -0.5 [-1.4 to 0.4] | -0.7 [-1.8 to 0.4]
  Week 4 (n=293, 144) | -0.5 [-1.5 to 0.5] | -1.0 [-2.1 to 0.2]
  Week 6 (n=280, 141) | -0.5 [-1.5 to 0.4] | -0.9 [-2.3 to 0.4]
  Week 8 (n=290, 142) | -0.0 [-1.0 to 1.0] | -0.7 [-2.0 to 0.6]
  Week 12 (n=286, 144) | 0.3 [-0.7 to 1.3] | 0.2 [-1.0 to 1.4]
  Week 16 (n=278, 139) | -1.0 [-2.1 to 0.1] | -0.6 [-2.1 to 1.0]
  Week 20 (n=276, 137) | -0.5 [-1.6 to 0.6] | 0.4 [-0.9 to 1.8]
  Week 24 (n=273, 134) | 0.0 [-1.2 to 1.3] | -1.0 [-2.5 to 0.4]
  Week 28 (n=264, 132) | -1.0 [-2.1 to 0.2] | -0.6 [-2.1 to 0.9]
  Week 36 (n=261, 129) | 0.0 [-1.1 to 1.2] | -0.0 [-1.4 to 1.4]
  Week 44 (n=250, 125) | 0.2 [-0.9 to 1.4] | -0.7 [-2.3 to 1.0]
  Week 52 (n=246, 125) | -0.3 [-1.5 to 0.8] | 0.2 [-1.7 to 2.1]

12. Other Pre Specified Outcome: Shift in Platelet Counts From Baseline to Selected Visits (LOCF)
Description: Platelet count=value*10^9 c/L
Time Frame: Baseline and Weeks 24 and 52
Population: All participants who received at least 1 dose of double-blind study medication.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 304 | 151
Participants
  Baseline <= 100; Week 24 <= 100 | 0 | 0
  Baseline <= 100; Week 24 >100 - <= 600 | 0 | 0
  Baseline <= 100; Week 24 >600 | 0 | 0
  Baseline >100 - <= 600; Week 24 <= 100 | 1 | 1
  Baseline >100 - <= 600; Week 24 >100 - <= 600 | 296 | 143
  Baseline >100 - <= 600; Week 24 >600 | 0 | 0
  Baseline >600; Week 24 <= 100 | 0 | 0
  Baseline >600; Week 24 >100 - <= 600 | 0 | 0
  Baseline >600; Week 24 >600 | 0 | 0
  Baseline <= 100; Week 52 <= 100 | 0 | 0
  Baseline <= 100; Week 52 >100 - <= 600 | 0 | 1
  Baseline <= 100; Week 52 >600 | 0 | 0
  Baseline >100 - <= 600; Week 52 <= 100 | 2 | 0
  Baseline >100 - <= 600; Week 52 >100 - <= 600 | 295 | 144
  Baseline >100 - <= 600; Week 52 >600 | 0 | 0
  Baseline >600; Week 52 <= 100 | 0 | 0
  Baseline >600; Week 52 >100 - <= 600 | 0 | 0
  Baseline >600; Week 52 >600 | 0 | 0

13. Other Pre Specified Outcome: Number of Participants With Marked Laboratory Abnormalities During the 24-Week ST + 52-Week LT Treatment Period
Description: Marked abnormality=a laboratory value lying outside the predefined criteria and more extreme (farther from the limit)on-treatment than at baseline. ULN=upper limit of normal; LLN=lower limit of normal; prx=pre-RX=pretreatment.
  Criteria 1: if prx=0 use >=2, if prx=0.5 or 1 use >=3, if prx=2 use 4.
Time Frame: Baseline and during and up to 14 days after last dose of study drug (in Week 52)
Population: All participants who received at least 1 dose of double-blind study medication.
Measure: Number; unit: Participants
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 304 | 151
Participants
  Hemoglobin <8 g/dL (n=300; 150) | 2 | 0
  Hematocrit <0.75*prx (n=300; 150) | 2 | 2
  Platelets <50*10^9 c/L (n=297; 145) | 0 | 0
  Platelets >1.5*ULN (n=297; 145) | 0 | 0
  Leukocytes <2*1000 c/uL (n=300; 150) | 0 | 1
  Neutrophils <1*1000 c/uL (n=296; 150) | 1 | 0
  Eosinophils >0.9*1000 c/uL (n=296; 150) | 9 | 7
  Lymphocytes <=0.75*1000 c/uL (n=296; 150) | 3 | 2
  Alkaline phosphatase >3*prx & >ULN (n=302; 150) | 2 | 1
  Alkaline phosphatase >1.5 ULN (n=302; 150) | 10 | 5
  Aspartate aminotransferase >3* ULN (n=298; 148) | 2 | 0
  Aspartate aminotransferase>5* ULN (n=298; 148) | 1 | 0
  Aspartate aminotransferase >10*ULN (n=298; 148) | 0 | 0
  Aspartate aminotransferase >20*ULN (n=298; 148) | 0 | 0
  Alanine transaminase >3*ULN (n=300; 148) | 5 | 3
  Alanine transaminase >5*ULN (n=300; 148) | 1 | 0
  Alanine transaminase >10*ULN (n=300; 148) | 0 | 0
  Alanine transaminase >20*ULN (n=300; 148) | 0 | 0
  Bilirubin, total >2 mg/dL (n=301; 150) | 0 | 0
  Bilirubin, total >1.5*ULN (n=301; 150) | 0 | 1
  Bilirubin, total >2*ULN (n=301; 150) | 0 | 0
  Blood urea nitrogen >2*prx & >ULN (n=302; 150) | 5 | 7
  Creatinine >2.5 mg/dL (n=303; 150) | 0 | 0
  Glucose, serum fasting <50 mg/dL (n=0; 0) | 0 | 0
  Glucose, serum fasting >500 mg/dL (n=0; 0) | 0 | 0
  Glucose, serum unspecified <50 mg/dL (n=0; 0) | 0 | 0
  Glucose, serum unspecified >500 mg/dL (n=0; 0) | 0 | 0
  Glucose, plasma fasting <50 mg/dL (n=301;150) | 5 | 0
  Glucose, plasma fasting >500 mg/dL (n=301;150) | 0 | 1
  Glucose, plasma unspecified <50 mg/dL (n=272; 133) | 5 | 1
  Glucose, plasma unspecified >500 mg/d (n=272; 133) | 1 | 1
  Sodium, serum <0.9*prx & <=130 mEq/L (n=302; 150) | 1 | 0
  Sodium, serum >1.1*prx & >=150 mEq/L (n=302; 150) | 0 | 0
  Potassium, serum <0.8 prx &<=3.2 mEq/L(n=300; 148) | 3 | 1
  Potassium, serum >1.2*prx&>= 6.0 mEq/L(n=300; 148) | 8 | 8
  Chloride, serum <90 mEq/L (n=302; 150) | 1 | 0
  Chloride, serum >120 mEq/L (n=302; 150) | 0 | 0
  Albumin <0.9*LLN; if prx<LLN, 0.75*prx (n=302,150) | 1 | 0
  Creatine kinase >5*ULN (n=301, 148) | 6 | 2
  Uric acid >1.5*ULN; if prx >ULN, >2 (n=0,0) | 0 | 0
  Protein urine (see criteria 1) (n=297,146) | 8 | 3
  Blood urine (see criteria 1) (n=297; 146) | 14 | 2
  Red blood cells urine (see criteria 1) (n=53; 31) | 8 | 3
  White blood cells urine (see criteria 1)(n=115;53) | 35 | 10

14. Other Pre Specified Outcome: Percentage of Participants With Reported and Confirmed Hypoglycemia
Description: Confirmed hypoglycemia=fingerstick glucose measurement of ≤50 mg/dL with associated symptoms/
Time Frame: Baseline to Week 52
Measure: Number; unit: Percentage of Participants
Arm/Group | Saxagliptin, 5 mg + Insulin | Placebo + Insulin
Number analyzed (Participants) | 300 | 149
Percentage of Participants
  Reported | 19.4 | 24.5
  Confirmed | 7.6 | 6.6

ADVERSE EVENTS:
Time Frame: Baseline to Week 52
Arm/Group | Placebo + Insulin | Saxagliptin, 5 mg + Insulin
Serious Adverse Events (participants affected / at risk) | 13/151 | 25/304
Other Adverse Events (participants affected / at risk) | 64/151 | 96/304
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Insulin (N=151) | Saxagliptin, 5 mg + Insulin (N=304)
DIABETIC RETINOPATHY (Eye disorders) | 0 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 1
CARDIAC FAILURE (Cardiac disorders) | 0 | 2
MYOCARDIAL ISCHAEMIA (Cardiac disorders) | 0 | 1
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 | 1
CORONARY ARTERY OCCLUSION (Cardiac disorders) | 0 | 1
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1
HYPERTENSION (Vascular disorders) | 0 | 1
PERIPHERAL ISCHAEMIA (Vascular disorders) | 1 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 1 | 0
THROMBOPHLEBITIS SUPERFICIAL (Vascular disorders) | 0 | 1
JAUNDICE (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS (Hepatobiliary disorders) | 1 | 0
CHOLANGITIS ACUTE (Hepatobiliary disorders) | 1 | 0
SCIATICA (Nervous system disorders) | 1 | 0
THALAMIC INFARCTION (Nervous system disorders) | 1 | 0
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 | 0
CONSTIPATION (Gastrointestinal disorders) | 0 | 1
CROHN'S DISEASE (Gastrointestinal disorders) | 0 | 1
PANCREATITIS CHRONIC (Gastrointestinal disorders) | 1 | 0
PNEUMONIA (Infections and infestations) | 0 | 1
BRONCHITIS (Infections and infestations) | 1 | 0
CELLULITIS (Infections and infestations) | 1 | 0
ABSCESS LIMB (Infections and infestations) | 2 | 0
DENGUE FEVER (Infections and infestations) | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 1 | 0
DIVERTICULITIS (Infections and infestations) | 0 | 1
ARTHRITIS INFECTIVE (Infections and infestations) | 1 | 0
INTESTINAL GANGRENE (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
RENAL IMPAIRMENT (Renal and urinary disorders) | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1 | 0
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
IRON DEFICIENCY ANAEMIA (Blood and lymphatic system disorders) | 1 | 0
ANAEMIA VITAMIN B12 DEFICIENCY (Blood and lymphatic system disorders) | 1 | 0
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 1 | 0
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 0
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 1 | 0
CHEST PAIN (General disorders) | 0 | 1
INFLUENZA LIKE ILLNESS (General disorders) | 1 | 0
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PITUITARY TUMOUR (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
UTERINE LEIOMYOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PANCREATIC CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PROSTATE CANCER METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo + Insulin (N=151) | Saxagliptin, 5 mg + Insulin (N=304)
HYPERTENSION (Vascular disorders) | 8 | 8
HEADACHE (Nervous system disorders) | 6 | 18
INFLUENZA (Infections and infestations) | 14 | 10
BRONCHITIS (Infections and infestations) | 4 | 16
PHARYNGITIS (Infections and infestations) | 8 | 11
NASOPHARYNGITIS (Infections and infestations) | 10 | 19
URINARY TRACT INFECTION (Infections and infestations) | 12 | 23
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 11 | 19
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 10 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication